CLINICAL TRIAL: NCT00217542
Title: A Phase 1 Study of 5-azacitidine in Combination With Interferon-Alfa 2B in Unresectable or Metastatic Melanoma and Renal Cell Carcinoma
Brief Title: Azacitidine and Recombinant Interferon Alfa-2b in Treating Patients With Stage III or Stage IV Melanoma or Stage IV Kidney Cancer That Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00152; YALE HIC#27409; YALE-HIC-27409; NCI-7317; CDR0000441640
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-05

CONDITIONS: Recurrent Melanoma; Recurrent Renal Cell Cancer; Stage III Melanoma; Stage IV Melanoma; Stage IV Renal Cell Cancer
MeSH Terms: conditions — Melanoma; Carcinoma, Renal Cell | interventions — Introns; Amifostine; Azacitidine

ARMS (1):
- Treatment (chemotherapy, biological therapy) (Experimental): Patients receive azacitidine SC once daily on days 1-4 and 15-17 and recombinant interferon alfa-2b SC on days 8, 10, 12, 15, 17, 19, 22, 24, and 26 during course 1. Beginning in course 2 and for all subsequent courses, patients receive azacitidine SC once daily on days 1-3 and 15-17 and interferon alfa-2b SC on days 1, 3, 5, 8, 10, 12, 15, 17, 19, 22, 24, and 26. Treatment repeats every 28 days for up to 12 total courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: recombinant interferon alfa-2b; Drug: amifostine/azacitidine

INTERVENTIONS:
Biological: recombinant interferon alfa-2b — Given SC
  Other Names: Alfatronol; Glucoferon; Heberon Alfa; IFN alpha-2B; Intron A
Drug: amifostine/azacitidine — Given SC

SUMMARY:
This phase I trial is studying the side effects and best dose of recombinant interferon alfa-2b when given together with azacitidine in treating patients with stage III or stage IV melanoma or stage IV kidney cancer that cannot be removed by surgery. Drugs used in chemotherapy, such as azacitidine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Recombinant interferon alfa-2b may interfere with the growth of tumor cells. Giving azacitidine together with recombinant interferon alfa-2b may kill more tumor cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the adverse event profile and maximum tolerated dose of interferon alfa-2b when combined with azacitidine in patients with unresectable stage III or IV melanoma or unresectable stage IV renal cell carcinoma.

II. Determine the feasibility of this regimen for future phase II trials.

OUTLINE: This is a dose-escalation, multicenter study.

Patients receive azacitidine subcutaneously (SC) once daily on days 1-4 and 15-17 and recombinant interferon alfa-2b SC on days 8, 10, 12, 15, 17, 19, 22, 24, and 26 during course 1. Beginning in course 2 and for all subsequent courses, patients receive azacitidine SC once daily on days 1-3 and 15-17 and interferon alfa-2b SC on days 1, 3, 5, 8, 10, 12, 15, 17, 19, 22, 24, and 26. Treatment repeats every 28 days for up to 12 total courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of interferon alfa-2b until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. After completion of study treatment, patients are followed every 2-4 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of 1 of the following:

  * Melanoma

    * Unresectable stage III disease
    * Stage IV disease
  * Renal cell carcinoma

    * Unresectable and/or stage IV disease
* Measurable disease
* No untreated brain metastases or leptomeningeal disease

  * Patients with previously treated brain metastases are eligible provided they have no evidence of progression for ≥ 4 weeks following treatment and do not require steroids
* Performance status - ECOG 0-2
* Performance status - Karnofsky 60-100%
* More than 3 months
* WBC ≥ 3,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9.0 g/dL (may be transfused to this level)
* PT or PTT < 1.5 times upper limit of normal (ULN)
* Bilirubin ≤ 2.0 mg/mL
* AST and ALT ≤ 3 times ULN (5 times ULN for patients with liver metastases)
* Albumin ≥ 3.0 g/dL
* Creatinine ≤ 1.7 mg/dL
* Creatinine clearance ≥ 50 mL/min
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No ventricular cardiac arrhythmia
* No myocardial infarction within the past 3 months
* No dyspnea at rest
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active gastrointestinal bleeding or ulcer disease
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study compliance
* No other uncontrolled illness
* No history of allergic reaction attributed to compounds of similar chemical or biologic composition to study agents
* At least 2 weeks since prior immunotherapy
* Prior adjuvant interferon alfa for metastatic disease or in the adjuvant setting allowed
* At least 3 weeks since prior cytotoxic agents (6 weeks for nitrosoureas or mitomycin)
* See Disease Characteristics
* At least 2 weeks since prior hormonal therapy
* At least 1 week since prior and no concurrent steroids
* At least 3 weeks since prior radiotherapy
* At least 2 weeks since prior minor surgery
* At least 3 weeks since prior major surgery
* Recovered from all prior therapy
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent investigational agents
* No other concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2005-07; Primary Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Adverse event profile of azacitidine and recombinant interferon alfa-2b in patients with unresectable or metastatic melanoma and renal cell carcinoma | Continuously throughout study
  Graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 3.0.
Maximum tolerated dose of recombinant interferon alfa-2b when administered in combination with 5-azacitidine | Course 1 (4 weeks)
  Toxicity will be graded according to the NCI CTCAE version 3.0. The MTD is the highest dose level in which < 2 patients of 6 develop first cycle DLT.
Correlation of promoter methylation with the level of expression of the genes | Day 5 or 8 and 24 or 26 of course 1
  Determined by Western blotting, immunohistochemistry, and/or RT-PCR. We will use Western blot analysis when antibodies are available and semi-quantitative RT-PCR in cases where antibodies are not available.

SECONDARY OUTCOMES:
Response rate of giving recombinant interferon alfa-2b when administered in combination with 5-azacitidine in patients with metastatic melanoma and renal cell carcinoma | Every 8 weeks
  Evaluated using the international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) Committee.

CONTACTS AND LOCATIONS:
Overall Officials: Mario Sznol, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States